CLINICAL TRIAL: NCT02189096
Title: Validation of Early Warning Score & Lactate in Prehospital Screening
Acronym: VELPS
Status: Completed | Type: Observational
Sponsor: University of the West of Scotland (Other)
Collaborators: Abbott Point of Care (Industry)
Responsible Party: Principal Investigator, Kevin Rooney, Professor, University of the West of Scotland
Other Study IDs: VELPS
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Sepsis
Keywords: Sepsis; National Early Warning Score; Lactate
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No change from current practice: Phase 1 (4 months)
  No change from current practice. Each Paramedic crew routinely documents patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be electronically captured. The data will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria [signs of systemic inflammation] and suspicion of infection) by the study investigators. An estimate will be made of the time of completion of the ePRF in relation to patient transport.
- NEWS and Sepsis Screening: Phase 2 (4 months)
  The ten crews will undertake implementation of NEWS and Sepsis Screening. Each Paramedic crew will continue to routinely document patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria and suspicion of infection). The NEWS will be available to the paramedic crew.
  If NEWS is greater than or equal to 4 or the patient screens positive for Sepsis, the patients transfer will be as per normal protocol but receiving ED staff will receive the information about NEWS score and Sepsis screening as part of a structured handover.
  Interventions: Other: NEWS and Sepsis Screening
- Point of care lactate measurement: Phase 3 ( 4 months)
  The ten crews will undertake Point of Care Lactate measurement when NEWS ≥ 4 or when the patient screens positive for Sepsis. Each Paramedic crew will continue to routinely document patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria and suspicion of infection).
  If NEWS is greater than or equal to 4 or the patient screens positive for Sepsis, then a Lactate will be measured on the CG4+ i-STAT cartridge. The lactate level, along with the NEWS score and sepsis screening, will be given to the receiving ED staff as part of a structured handover.
  Interventions: Other: Point of care lactate measurement

INTERVENTIONS:
Other: NEWS and Sepsis Screening — Each Paramedic crew will continue to routinely document patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria and suspicion of infection). The NEWS will be available to the paramedic crew.
  Groups: NEWS and Sepsis Screening
Other: Point of care lactate measurement — Each Paramedic crew will continue to routinely document patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria and suspicion of infection). If NEWS is greater than or equal to 4 or the patient screens positive for Sepsis, then a Lactate will be measured on the CG4+ i-STAT cartridge.
  Groups: Point of care lactate measurement

SUMMARY:
Sepsis claims over 37,000 lives in the United Kingdom each year- more than lung cancer, and more than breast cancer, bowel cancer and HIV/AIDS combined. Less than two-thirds of patients who develop sepsis will survive. Sepsis can affect a person of any age, social background, and can strike irrespective of underlying medical conditions.

An important element in improving the care of patient with sepsis is early identification and early intervention, both of which have been shown to improve outcomes. Physiological deterioration often precedes clinical deterioration as patients develop critical illness. Recognition of this has led to the development of Early Warning Score (EWS) systems which allow earlier identification of physiological deterioration. By assigning numerical values to various physiological parameters, a composite score can be assigned to a patient, allowing early identification of patients who are at risk of critical illness.

EWS were initially developed to assist in the management of patients in the general ward setting. A recent study has shown that an increased EWS on arrival at the Emergency Department (ED) is associated with higher odds of adverse outcome amongst patients with sepsis. Consequently, the use of EWS could facilitate patient pathways to ensure triage to a high acuity area of the ED and senior clinician involvement at an early stage. The use of a standard single National EWS (NEWS) across the National Health Service in the United Kingdom has been recommended to improve patient care.

NEWS also lends itself to extension to pre-hospital care and ambulance services. Most ambulance services routinely collect the physiological data required to calculate a NEWS score and indeed some ambulance services have incorporated this into electronic patient record forms (ePRF). An agreed NEWS score of greater than a specific level could be used as a trigger for ambulance service pre-alert of a receiving ED.

Point of care measurement of lactate has also been shown to be feasible in the ED. Serum lactate is recognised as an independent predictor of mortality in sepsis and there may be potential for combining NEWS systems and point of care to further improve diagnostic accuracy for patients at risk of adverse outcomes.

In this study, we aim to apply the use of early warning scores and point of care testing to a cohort of all ambulance patients to assess the feasibility and utility of this approach.

DETAILED DESCRIPTION:
Study Question or Objective:

Are NEWS score, Sepsis Screening and Lactate measurement predictors of outcome in unselected out of hospital patients?

Specific Aims:

To determine whether the following, alone or in combination, are predictors of outcome, namely in-hospital mortality within 24 hours or 30 days or ICU admission within two days:

* a single prehospital NEWS performed on arrival of the Scottish Ambulance Service (SAS)
* Prehospital Sepsis screening (SIRS criteria and evidence of infection) on arrival of the SAS
* Prehospital Point of Care Lactate performed when NEWS is greater than or equal to 4 or when Sepsis is present

Background Information:

NHS Scotland is committed to improving the outcome of patients with Sepsis and the Deteriorating Patient as evidenced by their inclusion in the Scottish Patient Safety Programme. An important element in improving the care of Sepsis and the deteriorating patient is early identification and early intervention, both of which have been shown to improve outcomes.

Physiological deterioration often precedes clinical deterioration as patients develop critical illness. Recognition of this has led to the development of Early Warning Scoring (EWS) systems, which allow earlier identification of physiological deterioration. By assigning numerical values to various physiological parameters, a composite score can be assigned to a patient, allowing early identification of patients who are at risk of critical illness.

EWS were initially established to assist in the management of patients in the general ward setting. A recent study has shown that an increased EWS on arrival at the Emergency Department (ED) is associated with higher odds of adverse outcome amongst patients with sepsis. Consequently, the use of EWS could facilitate patient pathways to ensure triage to a high acuity area of the ED and senior clinician involvement at an early stage. The use of a standard single National EWS (NEWS) across the National Health Service (NHS) in the United Kingdom has been recommended to improve patient care.

NEWS also lends itself to extension to prehospital care and ambulance services. Most ambulance services routinely collect the physiological data required to calculate a NEWS score and indeed some ambulance services have incorporated this into electronic patient report forms (ePRF). The Scottish Ambulance Service (SAS) has this in place. An agreed NEWS score of greater than a specific level could be used as a trigger for ambulance service pre-alert of a receiving ED. However controversy exists as to whether NEWS is valid in the prehospital environment.

Point of care lactate testing has also been shown to be feasible in the ED. Measurement of in hospital serum lactate is recognised as an independent predictor of mortality in sepsis and trauma and there may be potential for combining NEWS systems and point of care to further improve diagnostic accuracy for patients at risk of adverse outcomes. Prehospital Point of care lactate testing has also shown some promise as a predictor of outcome in trauma patients.

Previous studies have focused on using early warning scores and point of care lactate on specific patient groups. Identification of conditions such as sepsis can be challenging, particularly in the prehospital environment.

In this study, we aim to apply the use of early warning scores and point of care testing to a cohort of all ambulance patients to assess the feasibility and utility of this approach.

Study Design:

Setting Five areas within NHS Scotland have been identified and each area will have two paramedic crews taking part in the study. The five areas include NHS Greater Glasgow & Clyde (Royal Alexandra Hospital), NHS Dumfries & Galloway (Dumfries & Galloway Royal Infirmary), NHS Fife (Victoria Hospital), NHS Lothian (Royal Infirmary of Edinburgh) and NHS Western Isles (Western Isles Hospital). These areas have been chosen to represent the spectrum of clinical settings in NHS Scotland from dense urban areas to remote and rural area.

Posters will be placed in all ambulances in the five clinical areas informing patients that anonymised data is being collected for this study.

Methods The study will run for a 12-month period. The design is a prospective, non-randomised, 3 staged interventional study.

Phase 1 (4 months)

No change from current practice. Each Paramedic crew routinely documents patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be electronically captured. The data will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria [signs of systemic inflammation] and suspicion of infection) by the study investigators. An estimate will be made of the time of completion of the ePRF in relation to patient transport.

The National Early Warning Score (NEWS) contains seven physiological parameters, each of which is assigned a value of between 0 and 3 (0 and 2 for supplemental oxygen). The score for each parameter is summed to calculate the NEWS which may range between 0 and 20; the higher the score the greater the deviation from normality. The NEWS is based on previous similar scoring systems.

Sepsis is defined as the presence of SIRS criteria with the suspicion of infection.

Phase 2 (4 months)

The ten crews will undertake implementation of NEWS and Sepsis Screening. Prior to this stage of the study, each crew will attend a half day educational session covering the rationale for the use of NEWS.

Each Paramedic crew will continue to routinely document patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria and suspicion of infection). The NEWS will be available to the paramedic crew.

If NEWS is greater than or equal to 4 or the patient screens positive for Sepsis, the patients transfer will be as per normal protocol but receiving ED staff will receive the information about NEWS score and Sepsis screening as part of a structured handover.

Phase 3 ( 4 months)

The ten crews will undertake Point of Care Lactate measurement when NEWS ≥ 4 or when the patient screens positive for Sepsis. Each Paramedic crew will continue to routinely document patient observations in an electronic Patient Report Form (ePRF) on every patient encounter. These physiological parameters will be used to calculate NEWS and screen for Sepsis (2 or more modified SIRS criteria and suspicion of infection). If NEWS is greater than or equal to 4 or the patient screens positive for Sepsis, then a Lactate will be measured on the CG4+ i-STAT cartridge. The lactate level, along with the NEWS score and sepsis screening, will be given to the receiving ED staff as part of a structured handover.

Each crew will undergo a further half day educational session covering the use of the point of care lactate meter.

Within all NHS Scotland hospitals, health care practitioners currently screen for sepsis when NEWS is ≥ 4, and are measuring lactate if there is a positive screen for sepsis. Lactate point of care measurement is currently being piloted in the prehospital setting in Forth Valley Health Board

The i-STAT handheld analyser that will be used in this study is CE marked, and has undergone performance verification against GEM Premier 400 and ROCHE OMNI S blood gas analysers. It is currently used clinically within NHSGG&C health board, several other Scottish health boards and the Emergency Medical Retrieval Service (EMRS).

For the 12-month duration of the study paramedic crews will continue to work within Scottish Ambulance Service protocols and under the principles of UK Ambulance Clinical Practice Guidelines, including any changes made to SAS protocols during this time. Any changes will be noted by the study investigators.

Data Collection A researcher will obtain data for all patients in the study from the ePRF records via the SAS Data Warehouse. This data will be stored as a spreadsheet file in accordance with NHS data protection guidance. The researcher will then match this data with the Wardwatcher system at the receiving Intensive Care Units regarding ICU admission and ICU mortality. Data will be sought from <hospital information systems> at each receiving site regarding 30 day mortality.

Linked data will be anonymised and given a unique identifier. The anonymised data will then be analysed by an independent statistician, as described in the analysis plan.

Inclusion Criteria:

All patients attended to by these 10 paramedic teams over a 12-month period.

Exclusion Criteria:

Patients in cardiac arrest Children less than 16 years of age Patients with incomplete data collection

Primary Endpoint:

Primary endpoints are Intensive Care Unit (ICU) admission within 48 hours of attendance 24 hour mortality (all-cause) 30-day mortality (all cause, in hospital).

Secondary Endpoints:

Time from 999 call to ED arrival Time from Scottish Ambulance Service arrival to ED arrival (or first acute hospital assessment area) On-scene time for Scottish Ambulance Service Cost analysis

ELIGIBILITY:
Inclusion Criteria:

* All patients attended to by the assigned paramedic teams over a 12 month period

Exclusion Criteria:

* Patients in cardiac arrest
* Children less than 16 years of age
* Patients with incomplete data collection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from five Scottish healthboard areas.
Sampling Method: Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Intensive Care Unit admission within 48 hours of attendance | one year
  Intensive Care Unit admission within 48 hours of attendance 24 hour mortality (all cause) 30 day mortality (all cause, in hospital)

SECONDARY OUTCOMES:
Time from 999 call to ED arrival | one year
Time from Scottish Ambulance Service arrival to ED arrival | one year
On-scene time for Scottish Ambulance Service | one year
Cost analysis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Rooney, Principal Investigator — University of the West of Scotland